CLINICAL TRIAL: NCT05401019
Title: Efficacy of Treatment With Pramipexole or Risperidone in Patients With Refractory Obsessive-compulsive Disorder (OCD): Randomized Controlled Trial
Brief Title: Efficacy of Treatment With Pramipexole or Risperidone in Patients With Refractory Obsessive-compulsive Disorder (OCD)
Acronym: OCD-RT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This clinical trial was not approved by the regulatory entities. It was reviewed and a new trial was re-submitted.
Sponsor: Clinical Academic Center (2CA-Braga) (Other)
Collaborators: University of Minho (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OCD-RT; 2022-000249-34 (EudraCT Number)
Record Dates: First submitted 2022-05-25; First posted 2022-06-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-05

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Pramipexole; Risperidone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Treatment with pramipexol, once a day, tablet of 0.088, 0.18, 0.35, 0.53 mg per day during 16 weeks
  Interventions: Drug: Pramipexole
- Control arm (Active Comparator): Treatment with Risperidone, once a day, tablet of 0.5, 1, 1.5, 2 mg per day during 16 weeks + 8 weeks follow-up.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Pramipexole — Oral medication, once a day during 16 weeks
  Arms: Experimental arm
Drug: Risperidone — Oral medication, once a day during 16 weeks
  Arms: Control arm

SUMMARY:
This is a phase 2, randomized, controlled clinical trial to study the efficacy of pramipexol or risperidone in the treatment of refractory ODC patients.

This study is a two-parallel-group clinical trial with duration of 28 weeks (recruitment phase, 4 weeks + treatment phase, 16 weeks + follow-up phase, 8 weeks. The primary endpoint of this study is the score in the Y-BOCS scale measured between baseline and EOT ( at week 16).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 64 years;
2. European Portuguese as mother tongue;
3. Patients diagnosed with OCD, regardless of subtype, according to DSM-5 and/or ICD-10 criteria;
4. Yale-Brown Obsessive Compulsive Scale (Y-BOCS) score ≥ 16;
5. Patients who do not respond to treatment with at least two selective serotonin reuptake inhibitor antidepressants (SSRIs) at the maximum tolerated therapeutic dose with or without psychotherapy, i.e. patients in whom there is no reduction in the Y-BOCS score by 25% to 35% relative to the score obtained before starting treatment with SSRIs (Rauch & Jenike, 1994).

Exclusion Criteria:

1. Patients who have a complete response to drug treatment with or without psychotherapy, i.e. patients with a reduction in Y-Bocs score by 25% to 35% regarding the score obtained before starting treatment with SSRIS (Rauch & Jenike, 1994);
2. Patients with current or anterior history of psychotic illness (schizophrenia, delusions, among others);
3. Patients with bipolar disorder;
4. Patients with tick disorder;
5. Patients with borderline personality disorder;
6. Patients with social anxiety disorder;
7. Patients with current or anterior history of dietary behavior disorders (at least in the last 6 months);
8. patients with a history of neurological disease or traumatic brain injury;
9. Patients with history of alcohol abuse or illicit substances (at least in the last 6 months);
10. patients who are passing or have passed in the last 6 months by a major depressive episode;
11. Patients that undergo deep brain stimulation;
12. Presence of sensory deficits impeding participation in clinical study;
13. Pregnant or in breastfeeding period;
14. Patients doing medication or receiving prohibited treatments;
15. Patients with contraindication to perform MRI.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Y-BOCS total score | Change from Baseline Y-BOCS total score at visit 9 (16 weeks)
  Yale-Brown Obsessive Compulsive Scale (Y-BOCS) total score.
  The Y-BOCS scale measures obsessions separately from compulsions and specifically measures the severity of symptoms of obsessive-compulsive disorder without being biased towards or against the type of content the obsessions or compulsions might present.
  This instrument consists of 10 self-report items (5 items for obsessions, 5 items for compulsions) that estimate the degree of severity of symptoms (subclinical, mild, moderate, severe or extreme) on a Likert scale ranging from 0 (no symptoms) and 4 (extreme). The final score is calculated as the total sum of all items: subclinical (0 - 7 points), mild (8 - 15 points), moderate (16 - 23 points), severe (24-31) and extreme (32 - 40 points). In the final score, 16 is the cut-off point for symptom severity to be indicative of OCD

SECONDARY OUTCOMES:
Safety outcomes | Change from Baseline at visit 9 (16 weeks)
  Number of adverse events
Biochemical parameters | Change from Baseline at visit 9 (16 weeks)
  Complete blood count, cortisol, adrenocorticotropic hormone, thyroxine and thyroid stimulating hormone values
Neurobiological parameters | Change from Baseline at visit 9 (16 weeks)
  Cortical thickness; functional connectivity of neural networks and static and dynamic connectivity; brain activation during symptom induction; mean diffusivity, fractional anisotropy, axial diffusivity and radial diffusivity
Scores of the 4 subscales of the WHOQOL-bref | Change from Baseline at visit 9 (16 weeks)
  The Quality of Life Scale (WHOQOL-bref) is an instrument that assesses four conceptual domains of quality of life: material and physical well-being, relationships with other people, psychological well-being and environment.
  This self-report instrument, consisting of a brief sociodemographic questionnaire and 26 statements, quantifies global cognitive judgments of life satisfaction. The final score for each domain is calculated by adding up all the statements corresponding to that domain (D1: Physical - 7 items; D2: Psychological - 6 items; D3: Social Relations - 3 items; D4: Environment - 8 items).
OCI-R Total score | Change from Baseline at visit 9 (16 weeks)
  Obsessive-Compulsive Inventory-Revised (OCI-R) is an self-report instrument that assesses the symptoms of OCD during the last month through 18 statements that are related to everyday situations. The final score is calculated as the total sum of all items, ranging from 0 to 72, with a score greater than 20 indicative of severe symptoms of OCD.
PSS-10 Total score | Change from Baseline at visit 9 (16 weeks)
  Perceived Stress Scale (PSS-10) is a self-report questionnaire to assess perceived stress during the last month. The questionnaire's score is obtained by the sum of the answers in each item, which can vary between 0 and 40 points.
HAM-A Total score | Change from Baseline at visit 9 (16 weeks)
  Hamilton Anxiety Rating Scale (HAM-A) instrument to measure the psychic and somatic components of anxiety.
  The final score is calculated as the sum total of all items: mild anxiety (0 - 17 points), moderate anxiety (18 - 24 points) and potentially worrying levels of anxiety (25 - 30 points).
HAM-D Total score | Change from Baseline at visit 9 (16 weeks)
  Hamilton Depression Rating Scale (HAM-D) instrument to measure the psychic and somatic components of depression.
  The final score is calculated as the sum total of all items, from 0 - 7 the participant is considered asymptomatic, while a score equal to or greater than 20 indicates the presence of depressive symptoms. The higher the value, the greater the severity of the symptoms, ranging from moderate to severe.

IPD SHARING:
Plan to Share IPD: No